CLINICAL TRIAL: NCT02612467
Title: The Effectiveness of a Stratified Care Model for Non-specific Low Back Pain in Danish Primary Care Compared to Current Practice in a Randomised Controlled Trial
Brief Title: Low Back Pain - What's Next? Stratified Care Compared to Current Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: Herning Hospital (Other); Research Unit of General Practice, Odense (Other); Spine Centre of Southern Denmark (Other); Keele University (Other)
Responsible Party: Principal Investigator, Lars Morsoe, Ph.D., Region of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20140205
Record Dates: First submitted 2015-11-16; First posted 2015-11-23 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain
Keywords: start back tool; stratified care; targeted treatment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratified care (Experimental): Patients are stratified into low, medium, high risk of poor outcome. Stratified care are delivered by special trained physiotherapists according to risk group
  Interventions: Other: Stratified care
- Current care (Active Comparator): Treatment based on clinical judgement, clinical need and patient preferences. No access to guidance tools.
  Interventions: Other: Current care

INTERVENTIONS:
Other: Stratified care — Patients are stratified according to the SBT subgroups (low, medium and high risk) and the appropriate matched intervention will be delivered accordingly.
  Low risk: Reassuring information. Onwards referral, investigation or further treatment is not recommended Medium risk: In addition to reassuring information patients receive evidence based individualised treatment focusing on restoring function (targeting back pain, leg pain, co-morbid pain and disability) High risk : In addition to medium risk treatment patients will receive individualised psychologically informed physiotherapy aiming to reduce pain and disability.
  Arms: Stratified care
Other: Current care — Treatment based on clinical judgement, clinical need and patient preferences. No access to guidance tools.
  Arms: Current care

SUMMARY:
Background Studies in the United Kingdom find the stratified care model of the STarT Back Tool (SBT) to be superior to usual care in primary care low back pain (LBP) patients. However, considerations on differences in health care and social systems across countries are required before taking steps towards any recommendations of implementing stratified care into other health care services.

Objective To investigate the effectiveness of the stratified care model of the SBT, when embedded into the regional disease management programs on LBP in primary care as compared to current best practice care.

DETAILED DESCRIPTION:
Methods The study is a two-armed randomized controlled trial in Danish primary health care setting. In total 700 patients are included in the study.

The patients are randomised automatically by a developed database to; 1) Stratified care (treatment matched to stratification according to SBT) or 2) Control treatment (treatment based solely on clinical reasoning).

All data including patient consent is collected and monitored using a web-based data management system.

ELIGIBILITY:
Inclusion Criteria:

* patients found eligible for referral to physiotherapy by the general practitioner (GP)
* 18 years and above
* understand Danish language.

Exclusion Criteria:

* Serious pathology (malignancy, inflammatory arthritis, etc.),
* serious nerve root compression (cauda equina, paresis <3),
* influential comorbidity, psychiatric illness, personality disorder, spinal surgery during the last 6 months, pregnancy, or already receiving physiotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Patient reported change measured by the Roland Morris Disability Questionnaire | 3 and 12 months
  Change in disability measured by the Roland Morris Disability Questionnaire at 3 and 12 months (RMDQ)

SECONDARY OUTCOMES:
Cost-effectiveness across study arms measured by the EuroQol (EQ-5D) questionnaire | 12 months
  The health economic analysis will test the cost-effectiveness/cost-utility of SBT against current practice. Patient reported quality of life on the EuroQol (EQ-5D) questionnaire
Change in pain intensity measured on a numeric range scale | 3 and 12 months
  Change in pain intensity is monitored on numeric range scales indicating back and leg pain.
Time off work assessed by the Danish National Register on Public Transfer Payments (DREAM) | 3 and 12 months
  Short and long term time of work is monitored by standardized data from the Danish National Register on Public Transfer Payments (DREAM)
Time off work monitored by standardized patient reported data | 3 and 12 months
  Short and long term time of work is monitored by standardized patient reported data
Patient reported global change measured by the questionnaire "Global Impression of Change" | 3 and 12 months
  Patients perception of global change is monitored by the questionnaire "Global Impression of Change"

CONTACTS AND LOCATIONS:
Overall Officials: Lars Morsø, Ph.D, Principal Investigator — Centre for Quality, Institute for Regional Healthresearch
Locations (2):
- Denmark (2):
  - Department of Occ. Medicine, Herning, Central Region
  - Centre for Quality, Middelfart, Southern Denmark

REFERENCES:
- [Background] Morso L, Albert H, Kent P, Manniche C, Hill J. Translation and discriminative validation of the STarT Back Screening Tool into Danish. Eur Spine J. 2011 Dec;20(12):2166-73. doi: 10.1007/s00586-011-1911-6. Epub 2011 Jul 19. PMID 21769444
- [Result] Hill JC, Whitehurst DG, Lewis M, Bryan S, Dunn KM, Foster NE, Konstantinou K, Main CJ, Mason E, Somerville S, Sowden G, Vohora K, Hay EM. Comparison of stratified primary care management for low back pain with current best practice (STarT Back): a randomised controlled trial. Lancet. 2011 Oct 29;378(9802):1560-71. doi: 10.1016/S0140-6736(11)60937-9. Epub 2011 Sep 28. PMID 21963002
- [Derived] Morso L, Olsen Rose K, Schiottz-Christensen B, Sowden G, Sondergaard J, Christiansen DH. Effectiveness of stratified treatment for back pain in Danish primary care: A randomized controlled trial. Eur J Pain. 2021 Oct;25(9):2020-2038. doi: 10.1002/ejp.1818. Epub 2021 Jul 2. PMID 34101953
- [Derived] Morso L, Schiottz-Christensen B, Sondergaard J, Andersen NV, Pedersen F, Olsen KR, Jensen MS, Hill J, Christiansen DH. The effectiveness of a stratified care model for non-specific low back pain in Danish primary care compared to current practice: study protocol of a randomised controlled trial. Trials. 2018 Jun 8;19(1):315. doi: 10.1186/s13063-018-2685-5. PMID 29884217
- See also: Information regarding STarT Back Tool on the Keele University Homepage — http://www.keele.ac.uk/sbst/